CLINICAL TRIAL: NCT02073929
Title: A Randomised, Double-blind, Placebo-controlled Study of the Effect of Liraglutide in Polycystic Ovary Syndrome on Risk Markers of Vascular Thrombosis.
Brief Title: LIPT - Liraglutide in Polycystic Ovary Syndrome
Acronym: LIPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jens Faber (Other)
Responsible Party: Sponsor-Investigator, Jens Faber, Professor, DSc, Senior Hospital Physician, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT nr 2013-003862-15
Record Dates: First submitted 2014-02-25; First posted 2014-02-28 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2015-06

CONDITIONS: Polycystic Ovary Syndrome; Cardiovascular Disease
MeSH Terms: conditions — Polycystic Ovary Syndrome; Cardiovascular Diseases | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): Liraglutide s.c. 1,8mg daily for 26 weeks
  Interventions: Drug: Liraglutide for 26 weeks
- Placebo (Placebo Comparator): Placebo s.c. daily for 26 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Liraglutide for 26 weeks — GLP-1-analogue Liraglutide s.c. 1,8mg daily for 26 weeks
  Arms: Active
Drug: placebo — Placebo s.c. daily for 26 weeks
  Arms: Placebo

SUMMARY:
Polycystic ovary syndrome (PCOS) affects 5-10% of women in fertile age. PCOS is associated with metabolic syndrom, diabetes and and increased risk og cardiovascular disease.

The study investigates the effect af intervention with GLP-1-analog on risk markers of cardiovascular disease in women with PCOS.

70 women will be included in af RCT.

Hypothesis: GLP-1-analog treatment in women with PCOS (without diabetes) will result in a beneficial reduction in risk markers of vascular thrombosis and early cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* PCOS
* >18 years
* premenopausal
* BMI >25 og 25 and thereunder + insulin resistent

Exclusion Criteria (including):

* actualt or intended pregnancy
* inadeqvat contraception
* hormonal contraception within 6 weeks
* metfoomin, GLP-1-analog or DPP IV inhibitor within 3 months
* medications affectiv hemostatic mechanisme
* diabetes or other severe comorbidity
* familar MEN
* ...

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Faber, DSc, Principal Investigator — Dept. of Medicine, Herlev Hospital
Locations (3):
- Denmark (3):
  - Dept. of Medicine and Dept. of Gyn-Obs, Herlev Hospital, Herlev
  - Herlev Hospital, Dept of Gynecology, Herlev
  - Dept. of Medicine and Dept. of Obstetrics and Gynaecology, Herlev Hospital, Herlev

REFERENCES:
- [Derived] Frossing S, Nylander M, Chabanova E, Frystyk J, Holst JJ, Kistorp C, Skouby SO, Faber J. Effect of liraglutide on ectopic fat in polycystic ovary syndrome: A randomized clinical trial. Diabetes Obes Metab. 2018 Jan;20(1):215-218. doi: 10.1111/dom.13053. Epub 2017 Aug 11. PMID 28681988

RESULTS

PARTICIPANT FLOW:
Groups:
- Liraglutide: Liraglutide s.c. 1,8mg daily for 26 weeks
  Liraglutide: GLP-1-analogue Liraglutide
- Placebo: Placebo s.c. 1,8mg daily for 26 weeks
  placebo
Period: Overall Study
Arm/Group | Liraglutide | Placebo
Started | 48 | 24
Completed | 44 | 21
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Liraglutide: Liraglutide
- Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Placebo | Total
Number analyzed (Participants) | 48 | 24 | 72
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31.4 [24.6 to 35.6] | 26.2 [24.8 to 31.5] | 29.9 [24.7 to 34.2]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  women | 48 | 24 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  caucasians | 45 | 22 | 67
  other ethnicity | 3 | 2 | 5
BMI [Mean (Standard Deviation); unit: kg/m2] | 33.3 (5.1) | 33.3 (4.6) | 33.3 (4.9)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 102.6 (10.8) | 102.6 (11.1) | 102.6 (11.0)
Total testosterone [Median (Inter-Quartile Range); unit: nmol/l] | 1.23 [0.91 to 1.63] | 1.35 [0.95 to 1.93] | 1.30 [0.92 to 1.84]
Endogenous Thrombin Potential [Mean (Standard Deviation); unit: micromol/l x min] | 1796 (332) | 1830 (285) | 1801 (324)

OUTCOME MEASURES:

1. Primary Outcome: Change in Endogenous Thrombin Potential (ETP)
Description: Area under curve in a Thrombin Generation Test (TGT). Measurements every min for 10 min
Time Frame: at time 0 and 26 weeks
Measure: Mean (95% Confidence Interval); unit: nMolar x minutes
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 48 | 24
nMolar x minutes | -56.7 [-132.3 to 17.2] | -8.2 [-98.7 to 82.3]

2. Secondary Outcome: Percent Change in Plasma Level of Plasminogen Activator Inhibitor -1 PAI-1
Time Frame: at time 0 and 26 weeks
Measure: Mean (95% Confidence Interval); unit: percent change in plasma PAI-1
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 48 | 24
percent change in plasma PAI-1 | -12 [-23 to 0] | 4 [-14 to 26]

3. Other Pre Specified Outcome: Change in Plasma Level of Adrenomedullin
Description: measured in nmol/l
Time Frame: at time 0 and 26 weeks
Measure: Median (Inter-Quartile Range); unit: nmol/l
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 48 | 24
nmol/l | -0.02 [-0.04 to 0.002] | 0.003 [-0.02 to 0.02]

4. Other Pre Specified Outcome: Change in Plasma Level of Atrial Natriuretic Peptide (ANP)
Description: measured in pmol/l
Time Frame: at time 0 and 26 weeks
Measure: Median (Inter-Quartile Range); unit: pmol/l
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 48 | 24
pmol/l | -11.5 [-17.0 to -6.1] | 1.4 [-7.5 to 10.2]

5. Other Pre Specified Outcome: Change in Plasma Level of Copeptin
Time Frame: at time 0 and 26 weeks
Population: measured as pmol/l
Measure: Median (Full Range); unit: pmol/l
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 48 | 24
pmol/l | 0.48 [-0.39 to 1.34] | 0.28 [-0.51 to 1.08]

6. Other Pre Specified Outcome: Percent Change in Plasma Level of High Sensitivity C-reactive Protein (CRP)
Description: percent change from baseline
Time Frame: at time 0 and 26 weeks
Measure: Mean (Inter-Quartile Range); unit: percent change in CRP levels
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 48 | 24
percent change in CRP levels | -15 [-30 to 3] | -25 [-57 to 30]

7. Other Pre Specified Outcome: Change in Bleeding Pattern (Bleeding Ratio)
Description: Ration between number of bleedings during 3 months before trial and last 3 months of trial
Time Frame: at time 0 and 26 weeks
Measure: Median (Inter-Quartile Range); unit: n of bleedings/n of expected bleedings
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 48 | 24
n of bleedings/n of expected bleedings | 0.28 [0.20 to 0.36] | 0.14 [0.02 to 0.26]

8. Other Pre Specified Outcome: Change in Percent Liver Fat Content
Description: percent liver fat content
Time Frame: at time 0 and 26 weeks
Population: only participants with measurable i.e. >5% liver fat at baseline was included in this analysis
Measure: Mean (Standard Deviation); unit: percentage of liver fat
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 37 | 20
percentage of liver fat | -1.6 (0.4) | -0.2 (0.7)

9. Other Pre Specified Outcome: Change in Body Composition (VAT)
Description: cubic cm
Time Frame: at time 0 and 26 weeks
Population: not measured on all subjects (missing. 4 in Liraglutide and one in placebo Group)
Measure: Mean (Standard Deviation); unit: cubic cm
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 44 | 23
cubic cm | -17 (4) | 5 (7)

10. Other Pre Specified Outcome: Change in Ovarian Volume Between Baseline and Follow up (26 Weeks)
Description: measured as ml
Time Frame: at time 0 and 26 weeks
Population: not measured in all participants, one is missing in each group
Measure: Mean (95% Confidence Interval); unit: ml
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 47 | 23
ml | -2 [-3 to -1] | 0 [-2 to 1]

11. Other Pre Specified Outcome: Change in Serum Levels of Anti-Müllerian Hormone
Description: measured as pmol/l
Time Frame: at time 0 and 26 weeks
Population: missing one participant in placebo group
Measure: Mean (95% Confidence Interval); unit: pmol/ml
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 48 | 23
pmol/ml | -8.7 [-17.4 to 0.6] | 3.5 [-13.9 to 21.0]

ADVERSE EVENTS:
Groups:
- Active: Liraglutide s.c. 1,8mg daily for 26 weeks
  Liraglutide: GLP-1-analogue Liraglutide
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 2/48 | 1/24
Other Adverse Events (participants affected / at risk) | 37/48 | 3/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=48) | Placebo (N=24)
gallbladder stone attack (Hepatobiliary disorders) | 2 (2) | 1 (1) — gallbladder stone attack / gallstone related pain
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=48) | Placebo (N=24)
nausea (Gastrointestinal disorders) | 37 | 3 — nausea in up-titrating phase
constipation (Gastrointestinal disorders) | 12 | 0
vomiting (Gastrointestinal disorders) | 5 | 0
diarrhea (Gastrointestinal disorders) | 5 | 1
hypotension (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No